CLINICAL TRIAL: NCT01839227
Title: Post-operative Cognitive Dysfunction and the Change of Regional Cerebral Oxygen Saturation in Elderly Patients Undergoing Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1-2012-0039
Record Dates: First submitted 2013-04-16; First posted 2013-04-24 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Elderly Patients Undergoing Spinal Surgery
Keywords: Post-operative cognitive dysfunction; regional cerebral oxygen saturation; elderly
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- regional cerebral oxygen saturation (Experimental)
  Interventions: Other: Neurologic and neuropsychologic tests

INTERVENTIONS:
Other: Neurologic and neuropsychologic tests — Cognitive functioning was assessed with the following test: Korean Mini-Mental State Examination (K-MMSE) and visuomotor test of D-LOTCA battery.
  Regional cerebral oxygen saturation was continuously monitored using the INVOS 5100 (somatics,Troy, MI) with bifrontal placement of two sensors before the induction of the anesthesia until the end of operation.
  Baseline rSO2 was defined as the average saturation value over a 1 min period before induction of general anesthesia, beginning approximately 3 min after the sensors were applied in supine position. After the induction, baseline prone rSO2 was defined over a 5min period after the change of position.
  There is no intervention were made according to rSO2 values. Physiologic variables including BIS, PaCO2,PaO2, glucose, electrolyte, hematocrit, HR, MAP, and nasopharyngeal temperature were measured every 1 hours during the surgery.

SUMMARY:
Post operative cognitive dysfunction (POCD) is a well-recognized complication of patients undergoing cardiac surgery. Previous studies reported near-infrared spectroscopy provides information on the occurrence of cerebral desaturation resulted in POCD. But evidence of POCD after general surgery has been lacking. Especially, the prone position is used primarily for surgical access to the posterior spine, if there is any significant lowering of the legs or tilt of the entire table, venous returns may be decrease or augmented accordingly. The purpose of this study was to examine the relationship between POCD and intra-operative cerebral oxygen saturation after spine surgery in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* the patient undergoing the lumbar spine surgery in severance hospital

Exclusion Criteria:

* Patients who had previous cerebral disease, dementia, severe problems in hearing and understanding, or who were unable to provide informed consent were excluded.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
K-MMSE | change of K-MMSE from baseine to 1 month
  1. preoperative neuropsychological evaluation (the day before the surgery)
  2. intraoperative rSO2 data monitoring
  3-1. immediate postoperative neuropsychological evaluation (postoperative 4th~7th day)
  3-2. remote postoperative neuropsychological evaluation (postoperative 1month)
  4. Intraoperative

SECONDARY OUTCOMES:
visuomotor test(D-LOTCA battery) | measuring for visuomotor test during baseline and 1 month
  :Visuomotor test (D-LOTCA battery)
  * Copy Geometric Forms
  * Two Dimensional Model
  * Pegboard Construction
  * Block Design(colored)
  * Reproduction of Puzzle
  * Drawing Clock
Regional cerebral oxymetry monitoring | measuring for Regional cerebral oxymetry monitoring during baseline and 1 month
  * Correlation between rSO2 and POCD
    * The average, left and right absolute rSO2 values were collected every 30 seconds. rSO2 value was recorded as excel data.
    * Absolute rSO2 value and AUT(area under the threshold) send beneath the absolute threshold limits of 40%, 50%, 60% and 20% under the baseline. AUT was calculated based on this formula: AUT (present)=AUT (past)+(rSO2 threshold-rSO2 value)×sample rate
  * cutoff value of rSO2 predictive POCD
    * Correlation of physical value affecting rSO2 and POCD (BIS, PaCO2,PaO2, glucose, electrolyte, hematocrit, HR, MAP, and nasopharyngeal temperature, intraoperative blood loss, amount of intake fluid, total dose of vasopressor)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Annau Z. The effect of carbonic anhydrase inhibition on electrical self stimulation of the brain during hypoxia. Life Sci. 1977 Mar 15;20(6):1043-9. doi: 10.1016/0024-3205(77)90292-2. No abstract available. PMID 15172
- [Background] Cox PJ, Farmer PB, Jarman M, Kinas RW, Stec WJ. Stereoselectivity in the metabolism of the enantiomers of cyclophosphamide in mice, rats, and rabbits. Drug Metab Dispos. 1978 Nov-Dec;6(6):617-22. No abstract available. PMID 33022
- [Background] Stolke D, Seifert V. [Early or late operation on the ruptured aneurysm? An analysis based on 356 cases]. Neurochirurgia (Stuttg). 1988 May;31(3):81-7. doi: 10.1055/s-2008-1053907. German. PMID 3405354
- [Background] Al'tshuler NS. [Problems of tuberculosis control in the activities of the progressive medical community in prerevolutionary Russia]. Probl Tuberk. 1979 Dec;(12):62-5. No abstract available. Russian. PMID 392499
- [Background] Besch PK, Bermes EW Jr, McDonald HJ. Report of the second conference on education in clinical chemistry. Clin Chem. 1976 Apr;22(4):541-9. No abstract available. PMID 3299
- [Background] Tremblay NA, Davies DW, Volgyesi G, Kadar K, Steward DJ. Sodium nitroprusside: factors which attenuate its action. Studies with the isolated gracilis muscle of the dog. Can Anaesth Soc J. 1977 Nov;24(6):641-50. doi: 10.1007/BF03006708. PMID 22395
- [Background] Neutral all-purpose cleaner. Exec Housekeep Today. 1990 Nov;11(11):26. No abstract available. PMID 10107940
- [Background] Avolio G, Cacciabue M, Rolla G, Caria E, Oliaro A, Carlino F, Pepino E, Polizzi S, Bucca C. [Functional compromise of the small airways in subjects exposed to SiO2]. Minerva Med. 1986 Nov 30;77(45-46):2183-5. Italian. PMID 3025780
- [Background] Eulert J. [Transplantation of epiphyseal cartilage: experimental study]. Rev Chir Orthop Reparatrice Appar Mot. 1977;63 Suppl 2:136-7. No abstract available. French. PMID 143022
- [Background] Razin SV, Kekelidze MG, Lukanidin EM. [Spatial organization of replicons in the eukaryotic nucleus: attachment of replication initiation regions to the nuclear skeleton]. Mol Biol (Mosk). 1986 Mar-Apr;20(2):387-95. Russian. PMID 3010082
- [Background] Varki AP, Armitage JO, Feagler JR. Typhlitis in acute leukemia: successful treatment by early surgical intervention. Cancer. 1979 Feb;43(2):695-7. doi: 10.1002/1097-0142(197902)43:23.0.co;2-9. PMID 283878
- [Background] [Exosurf-Neonatal: the synthetic surfactant. Introductory symposium, 20 June 1992]. Monatsschr Kinderheilkd. 1992 Sep;140(9 [EXOSURF]):1-12. No abstract available. German. PMID 1406736
- [Background] Should I consider using an insulin pump to take insulin for type 2 diabetes? Johns Hopkins Med Lett Health After 50. 2004 Aug;17(6):8. No abstract available. PMID 15281175
- [Background] Kopacz DJ, Allen HW. Accidental intravenous levobupivacaine. Anesth Analg. 1999 Oct;89(4):1027-9. doi: 10.1097/00000539-199910000-00038. No abstract available. PMID 10512284
- [Background] Rossini F, Terruzzi E, Perego D, Miccolis I, Rivolta F, Manca E, Pogliani EM. Long-term follow-up of patients with intermediate or high-grade non-Hodgkin lymphoma treated with a combination of cyclophosphamide, epirubicin, vincristine, and prednisone. Cancer. 2004 Jan 15;100(2):350-5. doi: 10.1002/cncr.11907. PMID 14716771
- [Background] Panova MG, Sineshchekov VA, Karapetian NV. [Dependence of fluorescence spectra of chloroplasts from the activity of photosystem 2]. Mol Biol (Mosk). 1976 Sep-Oct;10(5):1175-82. Russian. PMID 1053077